CLINICAL TRIAL: NCT04425681
Title: Phase II Study of Osimertinib With Bevacizumab for Leptomeningeal Metastasis From EGFR-mutation Non-Small Cell Lung Cancer
Brief Title: Osimertinib With Bevacizumab for Leptomeningeal Metastasis From EGFR-mutation Non-Small Cell Lung Cancer
Acronym: OWBLM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20161BBG70210
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Leptomeningeal Metastasis; Non-small Cell Lung Cancer; EGFR Activating Mutation
Keywords: leptomeningeal metastasis; non small cell lung cancer; EGFR Activating Mutation; Osimertinib; Bevacizumab
MeSH Terms: conditions — Meningeal Carcinomatosis; Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib With Bevacizumab group (Experimental): Osimertinib 80 mg oral daily; and bevacizumab 7.5 mg/kg intravenous every 3 weeks
  Interventions: Drug: Osimertinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Osimertinib — Treatment of LM With osimertinb
Drug: Bevacizumab — Treatment of LM With Bevacizumab

SUMMARY:
Leptomeningeal metastasis (LM) is a fatal complication of advanced non-small cell lung cancer (NSCLC) associated with poor prognosis and rapid deterioration of performance status. The incidence of LM is increasing, reaching 3.8% in molecularly unselected NSCLC patients, being more frequent in adenocarcinoma subtype and up to 9% in epidermal growth factor receptor mutation (EGFRm) lung cancer patients, one-third of patients have concomitant brain metastasis . This increased incidence may in part be conducive to the increased survival of patients with EGFRm advanced NSCLC since the introduction of EGFR-tyrosine kinase inhibitions (TKIs).Currently, no standard therapeutic regimen for LM has been established because of its rarity and heterogeneity[11], and no approved therapies exists to specifically target LM in patients with EGFRm NSCLC. TKIs therapy is the first-line treatment of patients with EGFRm of NSCLC. The leptomeningeal space is a sanctuary site for tumour cells and therapeutic agents due to the presence of an active blood-brain barrier (BBB), so CSF concentration is an important factor affecting treatment of LM by TKIs. Standard-dose first- and second-generation EGFR-TKIs have good systemic efficacy but sub-optimal CNS penetration, as evidenced by preclinical studies of brain distribution and clinical reports of CSF penetration[15, 16]. Osimertinib is a third-generation EGFR-TKI, irreversible, oral EGFR-TKI that potently and selectively inhibits both EGFR-TKI sensitizing and EGFR T790M resistance mutations, which has demonstrated efficacy in NSCLC CNS metastasis[17-22]. Preclinical, I/II clinical studies and AURA program (AURA extension, AURA2, AURA17 and AURA3) have shown that Osimertinib has higher brain permeability than the first- and second-generation.

Bevacizumab is a recombinant humanized monoclonal antibody against vascular endothelial growth factor (VEGF), animal studies and autopsy specimens show that VEGF plays an important role in LM. VEGF and EGFR share many overlapping and parallel downstream pathways. The biological rationale shows that inhibiting of EGFR and VEGR signaling pathways could improve the efficacy of antitumor and remove the resistance of EGFR inhibition. Besides, preclinical researches have shown the similar results. Based on these, numbers of clinical trials have confirmed that VEGF inhibitors in combination with EGFR-TKI significantly prolong patients' survival.

DETAILED DESCRIPTION:
This is a phase II pilot study to evaluate the efficacy and safety of osimertinib with bevacizumab for LM from EGFRm NSCLC patients. ALL patients were treated with Osimertinib 80mg oral daily and bevacizumab 7.5mg/kg intravenous every 3 weeks. Study therapy continued until disease progression, unacceptable adverse event, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Age in 18-80 years
* Pathologically proven NSCLC
* EGFR mutation , the EGFR status was identified from primary lung tumors using the amplification refractory mutation system (ARMS) or next-generation sequencing (NGS) analysis.
* LM diagnosis was based on the detection of malignant cells in the CSF, the focal or diffuse enhancement of leptomeninges, and nerve roots or the ependymal surface on gadolinium-enhanced MRI .
* No severe abnormal liver and kidney function;
* No other severe chronic diseases;
* Signed informed consent form

Exclusion Criteria:

* Patients with the clinical manifestation of nervous system failure including severe encephalopathy, grade III-IV white matter lesions confirmed by imaging examination, moderate or severe coma, and glasgow coma score less than 9 points;
* Allergic to osimertinib or bevacizumab
* Any of the following: Pregnant women ;Nursing women ;Men or women of childbearing potential who are unwilling to employ adequate contraception
* History of myocardial infarction or other evidence of arterial thrombotic disease (angina), symptomatic congestive heart failure (New York Heart Association ≥ grade 2), unstable angina pectoris, or cardiac arrhythmia; Note: allowed only if patient has no evidence of active disease for at least 6 months prior to randomization;
* History of cerebral vascular accident (CVA) or transient ischemic attack (TIA)≤ 6 months prior to randomization
* History of bleeding diathesis or coagulopathy
* History of hemoptysis da≥ grade 2 (defined as bright red blood of at least 2.5 mL) ≤3 months prior to randomization
* Leukocytes below 2*10^9/L, neutrophils below 1*10^9/L; platelets below 50*10^9/L;
* Had major surgery within 60 days;
* History of arteriovenous thrombosis
* Gastrointestinal perforator in the past 6 months
* Inadequately controlled hypertension (systolic blood pressure of > 150 mmHg or diastolic pressure > 100 mmHg on anti-hypertensive medications); Note: history of hypertensive crisis or hypertensive encephalopathy not allowed
* Grade 4 proteinuria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
LM progression-free survival | up to 1 year
  Time from LM diagnosis to the first documentation of disease progression or death
Objective Response Rate | up to 1 year
  ORR, proportion of patients with a best overall response of complete response or partial response (CR+PR)

SECONDARY OUTCOMES:
LM Overall survival | Every 6 weeks, up to 2 years
  LM-OS defined as time from LM diagnosis to death due to any cause or last follow-up
progression-free survival | Every 6 weeks, up to 2 years
  Proportion of patients progression-free by investigator assessment per RECIST v1.1
adverse events | Every 3 weeks, up to 2 years
  Number of patients with adverse events (AEs) as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Liu Anwen, Phd, Study Director — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Afiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramalingam SS, Vansteenkiste J, Planchard D, Cho BC, Gray JE, Ohe Y, Zhou C, Reungwetwattana T, Cheng Y, Chewaskulyong B, Shah R, Cobo M, Lee KH, Cheema P, Tiseo M, John T, Lin MC, Imamura F, Kurata T, Todd A, Hodge R, Saggese M, Rukazenkov Y, Soria JC; FLAURA Investigators. Overall Survival with Osimertinib in Untreated, EGFR-Mutated Advanced NSCLC. N Engl J Med. 2020 Jan 2;382(1):41-50. doi: 10.1056/NEJMoa1913662. Epub 2019 Nov 21. PMID 31751012
- [Result] Flippot R, Biondani P, Auclin E, Xiao D, Hendriks L, Le Rhun E, Leduc C, Beau-Faller M, Gervais R, Remon J, Adam J, Planchard D, Lavaud P, Naltet C, Caramella C, Le Pechoux C, Lacroix L, Gazzah A, Mezquita L, Besse B. Activity of EGFR Tyrosine Kinase Inhibitors in NSCLC With Refractory Leptomeningeal Metastases. J Thorac Oncol. 2019 Aug;14(8):1400-1407. doi: 10.1016/j.jtho.2019.05.007. Epub 2019 May 18. PMID 31108248
- [Result] Akamatsu H, Teraoka S, Morita S, Katakami N, Tachihara M, Daga H, Yamamoto N, Nakagawa K. Phase I/II Study of Osimertinib With Bevacizumab in EGFR-mutated, T790M-positive Patients With Progressed EGFR-TKIs: West Japan Oncology Group 8715L (WJOG8715L). Clin Lung Cancer. 2019 Jul;20(4):e492-e494. doi: 10.1016/j.cllc.2019.03.002. Epub 2019 Mar 19. PMID 31085043
- [Result] Wu YL, Ahn MJ, Garassino MC, Han JY, Katakami N, Kim HR, Hodge R, Kaur P, Brown AP, Ghiorghiu D, Papadimitrakopoulou VA, Mok TSK. CNS Efficacy of Osimertinib in Patients With T790M-Positive Advanced Non-Small-Cell Lung Cancer: Data From a Randomized Phase III Trial (AURA3). J Clin Oncol. 2018 Sep 10;36(26):2702-2709. doi: 10.1200/JCO.2018.77.9363. Epub 2018 Jul 30. PMID 30059262
- [Result] Taillibert S, Chamberlain MC. Leptomeningeal metastasis. Handb Clin Neurol. 2018;149:169-204. doi: 10.1016/B978-0-12-811161-1.00013-X. PMID 29307353
- [Result] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359
- [Result] Gregorc V, Lazzari C, Karachaliou N, Rosell R, Santarpia M. Osimertinib in untreated epidermal growth factor receptor (EGFR)-mutated advanced non-small cell lung cancer. Transl Lung Cancer Res. 2018 Apr;7(Suppl 2):S165-S170. doi: 10.21037/tlcr.2018.03.19. No abstract available. PMID 29782558
- [Result] Cross DA, Ashton SE, Ghiorghiu S, Eberlein C, Nebhan CA, Spitzler PJ, Orme JP, Finlay MR, Ward RA, Mellor MJ, Hughes G, Rahi A, Jacobs VN, Red Brewer M, Ichihara E, Sun J, Jin H, Ballard P, Al-Kadhimi K, Rowlinson R, Klinowska T, Richmond GH, Cantarini M, Kim DW, Ranson MR, Pao W. AZD9291, an irreversible EGFR TKI, overcomes T790M-mediated resistance to EGFR inhibitors in lung cancer. Cancer Discov. 2014 Sep;4(9):1046-61. doi: 10.1158/2159-8290.CD-14-0337. Epub 2014 Jun 3. PMID 24893891
- [Result] Umemura S, Tsubouchi K, Yoshioka H, Hotta K, Takigawa N, Fujiwara K, Horita N, Segawa Y, Hamada N, Takata I, Yamane H, Kamei H, Kiura K, Tanimoto M. Clinical outcome in patients with leptomeningeal metastasis from non-small cell lung cancer: Okayama Lung Cancer Study Group. Lung Cancer. 2012 Jul;77(1):134-9. doi: 10.1016/j.lungcan.2012.03.002. Epub 2012 Apr 7. PMID 22487432
- [Result] Tabernero J. The role of VEGF and EGFR inhibition: implications for combining anti-VEGF and anti-EGFR agents. Mol Cancer Res. 2007 Mar;5(3):203-20. doi: 10.1158/1541-7786.MCR-06-0404. PMID 17374728
- [Result] De Luca A, Carotenuto A, Rachiglio A, Gallo M, Maiello MR, Aldinucci D, Pinto A, Normanno N. The role of the EGFR signaling in tumor microenvironment. J Cell Physiol. 2008 Mar;214(3):559-67. doi: 10.1002/jcp.21260. PMID 17894407
- [Result] Lv Y, Mu N, Ma C, Jiang R, Wu Q, Li J, Wang B, Sun L. Detection value of tumor cells in cerebrospinal fluid in the diagnosis of meningeal metastasis from lung cancer by immuno-FISH technology. Oncol Lett. 2016 Dec;12(6):5080-5084. doi: 10.3892/ol.2016.5314. Epub 2016 Oct 25. PMID 28105214
- [Result] Hochmair M. Medical Treatment Options for Patients with Epidermal Growth Factor Receptor Mutation-Positive Non-Small Cell Lung Cancer Suffering from Brain Metastases and/or Leptomeningeal Disease. Target Oncol. 2018 Jun;13(3):269-285. doi: 10.1007/s11523-018-0566-1. PMID 29700687
- [Result] Masuda C, Yanagisawa M, Yorozu K, Kurasawa M, Furugaki K, Ishikura N, Iwai T, Sugimoto M, Yamamoto K. Bevacizumab counteracts VEGF-dependent resistance to erlotinib in an EGFR-mutated NSCLC xenograft model. Int J Oncol. 2017 Aug;51(2):425-434. doi: 10.3892/ijo.2017.4036. Epub 2017 Jun 8. PMID 28627678